CLINICAL TRIAL: NCT03740906
Title: Direct-acting Antiviral Therapy and Reinfection Among People With Chronic Hepatitis C Virus Infection and Recent Injecting Drug Use in the Prison Setting (The SHARP-P Study)
Brief Title: Direct-acting Antiviral Therapy and Reinfection Among People With Chronic Hepatitis C Virus Infection and Recent Injecting Drug Use in the Prison Setting
Acronym: SHARP-P
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHCRP1606
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Plasma, PBMCs, Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SHARP-P is an observational cohort study investigating the effect of direct-acting antiviral (DAA) therapy and reinfection in people with chronic hepatitis C virus (HCV) and recent injecting drug use. A prospective, observational cohort design will be used to enrol patients from correctional centres in New South Wales, Australia.

Participants will be prescribed a direct-acting HCV medication as per the standard of care. The on treatment phase will vary dependent on the type of a direct-acting antiviral prescribed as per the standard of care. Once patients have completed their treatment course they will be followed up every 3 months for up to 3 years following the end of treatment phase.

The study will aim to evaluate the incidence of HCV reinfection following successful DAA treatment over the three years of follow up. The study will also evaluate the proportion of patients with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) with direct-acting anti-viral HCV therapy.

DETAILED DESCRIPTION:
In Australia, hepatitis C virus (HCV)-related morbidity and mortality have doubled in the past decade, with health care costs of $220 million per annum associated with approximately 200,000 chronically infected cases. The majority of new (90%) and existing (80%) cases of HCV infection occur among people who inject drugs (PWID).

As there is a close relationship between imprisonment, injecting drug use, and HCV, in any given year, almost 20,000 of those with chronic HCV in Australia spend time in prison, including approximately 8,000 in New South Wales (NSW). These individuals are likely to represent the most marginalised and 'hard-to-access' subgroup of the affected population. In addition, the prison environment is a key venue for ongoing transmission. Amongst PWID in the prison setting the report of any injecting drug use decreased from 71% prior to prison entry to 27% following imprisonment. However, among people who reported injecting drug use, the proportion reporting sharing a needle/syringe increased from 29% prior to prison entry to 73%. In the community, 15-20% of current PWID report recent (last month) receptive needle/syringe sharing.

In prison, where there is no access to formal needle and syringe programs, sharing injecting equipment can be normative with inmates' accounts of injecting practice revealing few ways that they can minimise HCV risk. Establishing effective disease prevention in the prison context is challenging, as prisons are unique in physical structure, and prisoners form a distinct micro-society with their own rules and regulations. Many health problems amongst prisoners arise directly from conditions of imprisonment such as overcrowding, uncontrolled exposure to violence and illicit drugs, lack of purposeful activity, separation from family networks and emotional deprivation.

The existing strategies for HCV prevention in NSW prisons are delivered by Justice Health & Forensic Mental Health and Corrective Services. Justice Health & Forensic Mental Health provides a targeted screening program for blood-borne virus infection with pre- and post-test counselling, and opioid substitution treatment (OST) for those who are opioid dependent. Corrective Services provides bleach (or the quaternary amine disinfectant, Fincol) to clean used syringes. NSP is not available.

Despite these efforts, in the Hepatitis C Incidence and Transmission Study in prisons (HITS-p; n=590) led by CI-Lloyd, half of the cohort (49%) of PWID reported injecting drug use during follow-up in prison and 31% reported sharing injecting equipment. HCV incidence was 14.1/100 p-yrs (95% CI: 9.96, 19.3). There was no apparent protective effect of bleach cleansing or OST, highlighting the additional challenges of HCV prevention in the custodial setting.

Qualitative research shows that decisions about sharing equipment are multi-factorial and can include issues ranging from service access (such as distance to service and opening hours), concerns about anonymity, perceptions that HCV is ubiquitous and unavoidable to socially-located concerns that promote use of sterile equipment such as a desire to avoid "track marks". In the prison context, complex social, economic, and environmental risk factors contributed to injecting practices with the person supplying the drugs injecting first, and the person who owns the injecting equipment going next. Risk of HCV acquisition did not regularly factor into determining order of injection within networks. There is no research that examines sharing of injecting equipment in those who have been cured with antiviral therapy in either community or prison settings.

Increasing access to HCV therapy is a key objective of national and NSW Hepatitis C Strategies. The advent of well-tolerated, simple, oral hepatitis C virus (HCV) regimens - direct acting antivirals (DAAs) - has the potential to transform this landscape. These are much shorter, tolerable treatment regimens with cure rates >95%, providing an opportunity to reverse the rising burden of advanced liver disease. From 1st March 2016, these highly efficacious HCV therapies have been listed on the Pharmaceutical Benefit Scheme, and people with recent injecting drug use including prisoners are eligible to receive them. These are important features of the listing. In many countries, people who have not ceased injecting drug use are ineligible to receive DAA therapy, despite the fact that they comprise a significant proportion of HCV cases. Australia is therefore is leading the world in the scale-up of new therapies to an extent that many countries with such exclusions will not be able to achieve.

This feature of DAA access also affords unique opportunities with respect to the implementation of treatment scale-up in community drug treatment clinics and prisons. Australia has good treatment coverage for people who are opioid dependent, with over 50% of opioid dependent people estimated to engage in opioid substitution therapy (OST). Community-based drug treatment clinics and prisons represent a logical venue for expansion of HCV care beyond existing tertiary HCV treatment centres.

Although response to DAA HCV therapy is high, lower responses have been observed among people with previous treatment experience, cirrhosis and those with baseline or emergent resistance associated variants. Such resistance associated variants can persist for up to two years after treatment, affect re-treatment options, and be transmitted to new hosts. Further, PWID are likely to be exposed to multiple HCV infections as a result of ongoing high-risk behaviours and might commonly harbour mixed HCV infections (infection with two or more distinct viruses). Underlying mixed HCV infection can contribute to nonresponse during therapy, which has implications for DAA regimens that are preferentially active against specific viral genotypes or subtypes. These data argue for surveillance of HCV resistance and mixed HCV infection among PWID to resolve residual concerns regarding their clinical and public health significance.

Two systematic reviews assessing interferon-based therapy for PWID have demonstrated responses comparable to randomised controlled trials excluding PWID. These data have supported international recommendations for the management of HCV for PWID. However, there are limited data on DAA therapy among recent PWID. As treatment is broadened to include more marginalised individuals, many clinicians are reluctant to treat HCV among PWID with recent injecting drug use with new DAA therapies. Major concerns include poor adherence/response, increased risk behaviour and HCV reinfection.

A major concern is that ongoing injecting risk behaviours following DAA therapy in PWID will lead to HCV reinfection, reversing the benefits of cure. Ongoing risk behaviours following successful HCV therapy may lead to reinfection and compromised treatment outcomes. In a systematic review and meta-analysis of HCV reinfection among PWID performed by the investigators, the pooled estimate of re-infection was 2.2/100 p-yrs (95% CI, 0.9-6.1) overall and 6.4/100 p-yrs (95% CI, 2.5-16.7) among individuals who reported injecting drug use post-SVR. The one study of HCV reinfection post-therapy in prison performed to date was small (n=74), retrospective, and did not assess the rate of HCV reinfection. Studies of reinfection following HCV therapy are limited by small sample sizes, retrospective study designs, incomplete follow-up, and a lack of sensitive methods to detect reinfection. Further, there are no data on HCV reinfection among recent PWID treated with DAAs.

Although DAA therapy could limit HCV-related disease burden, as treatment is broadened to include more marginalised individuals, many clinicians are reluctant to treat HCV among recent PWID, given concerns about poor adherence (and lower response to therapy), increased risk behaviours (due to the ease and high cure rates of DAA HCV therapy) and HCV reinfection (thereby reversing cure). However, no data exist on the extent to which this should be a concern. Given that DAA HCV therapy is highly expensive, we urgently need data on the magnitude of risk for, and predictors of, HCV reinfection. It is also unclear whether PWID treated in these two settings will vary in their response to DAA therapy and risk for reinfection.

The investigators have an excellent track record of conducting high quality cohort studies and clinical trials among PWID in the community and prison, with high participant retention in follow-up. The investigators have developed a network of community-based clinical sites providing HCV care in nine community-based drug treatment clinics, and many years of collaborative clinical research in the prison sector. In SHARP the investigators will explore the risk of HCV reinfection and treatment efficacy among recent PWID with chronic HCV and recent injecting drug use in the community and in the prisons.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have voluntarily signed the informed consent form.
2. Be ≥18 years of age on day of signing informed consent form.
3. Have chronic HCV infection.
4. Report of recent injecting drug use (within the previous 6 months).
5. Eligible for DAA therapy as per the PBS
6. HIV-1 infected participants enrolled in the study must meet the following additional criteria:

   1. Have HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry (Baseline) and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load.
   2. Be on HIV Antiretroviral Therapy (ART) for at least 4 weeks prior to study entry using an ART regimen that is allowable with the intended DAA regimen as determined by the current PI and the Liverpool drug interaction website (http://www.hiv-druginteractions.org/) OR be naive to treatment with any antiretroviral therapy (ART) with a baseline CD4 count of >200 and have no plans to initiate ART treatment while participating in this study and through to at least Follow-up Week 4.

Exclusion Criteria:

1. The participant will be excluded from participating in the study if the subject is unable or unwilling to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with chronic HCV infection and recent injecting drug use who are 18 years or over and are eligible for DAA therapy as per the PBS criteria
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of HCV reinfection following successful DAA therapy among people with chronic HCV infection and recent injecting drug use in the prison setting. | 3 years

SECONDARY OUTCOMES:
To evaluate the proportion of participants with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) following DAA HCV therapy among PWID with chronic HCV infection and recent injecting drug use | 2.5 years
To evaluate the proportion of participants who complete treatment | 3 years
To evaluate the proportion of participants with undetectable HCV RNA at the end of treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lloyd, Principal Investigator — Kirby Institute
Locations (1):
- NSW Correctional Centres, Sydney, New South Wales, Australia